CLINICAL TRIAL: NCT02270554
Title: A Prospective, Multi-center Investigation of Impact of the Endo GIA Reinforced Reload With Tri-Staple Technology During Distal Pancreatectomy
Brief Title: A Prospective, Multi-center Trial for Reinforced Staple During Distal Pancreatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wakayama Medical University (Other)
Responsible Party: Principal Investigator, Hiroki Yamaue, Second Deaprtment of Surgery, Wakayama Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DP-Study 1401
Record Dates: First submitted 2014-10-10; First posted 2014-10-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Reinforced staple (Experimental): Endo GIA Reinforced Reload with Tri-Staple technology
  Interventions: Device: Endo GIA Reinforced Reload with Tri-Staple technology

INTERVENTIONS:
Device: Endo GIA Reinforced Reload with Tri-Staple technology — Device:Endo GIA Reinforced Reload with Tri-Staple technology

SUMMARY:
The aim of this study is to evaluate if the Endo GIA Reinforced Reload with Tri-Staple Technology reduce incidence of pancreatic fistula (ISGPF grade B and C) after distal pancreatectomy by a prospective, multi-center trial.

DETAILED DESCRIPTION:
Reducing the incidence of pancreatic fistula is the most important issue in pancreatectomy. There is no certain view on the pancreatic resection method to reduce pancreatic fistula in distal pancreatectomy.This study will be conducted to scientifically investigate the impact of Endo GIA Reinforced Reload with Tri-Staple Technology in distal pancreatectomy. The aim of this study is to evaluate if the Endo GIA Reinforced Reload with Tri-Staple Technology reduce incidence of pancreatic fistula (ISGPF grade B and C) after distal pancreatectomy by a prospective, multi-center trial.

ELIGIBILITY:
Inclusion Criteria:

1. disease of pancreatic body and tail
2. PS (ECOG Performance Status Scale)0-1
3. Age: 20 years or older
4. distant metastases are not diagnosed preoperatively. Eligible for this clinical study when only distal pancreatectomy contributes to the favorable prognosis even if patients with pancreatic neuroendocrine cancer have the liver metastasis
5. Patients who can provide written informed consent

Exclusion Criteria:

1. Patients with severe ischemic cardiac disease
2. Patients with severe liver cirrhosis or active hepatitis
3. Patients with respiratory illness that requires oxygen administration
4. Patients with chronic renal failure requiring dialysis
5. Patients requiring other organ resection
6. Patients who are unfit for the study as determined by the attending physician

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Incidence of pancreatic fistula grade B/C | Ninety days after operation

SECONDARY OUTCOMES:
Incidence of pancreatic fistula defined by ISGPF classification | Ninety days after operation
Incidence of pancreatic fistula grade C defined by ISGPF classification | Ninety days after operation
Incidence of intraabdominal bleeding | Ninety days after operation
Morbidity | Ninety days after operation
Mortality | Ninety days after operation
Postoperative hospital stay | Ninety days after operation
Hemostasis condition of staple line | during operation
Malformationof staple line Malformationof staple line Malformationof staple line Malformationof staple line Malformationof staple line | during operation
Period of drain insertion | Ninety days after operation
Damage of pancreatic stump | during operation
Frequency of additional suture of pancreatic stump | during operation
Incidence of pancreatic fistula stratified based on thickness of pancreas parenchyma | Ninety days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Hiroki Yamaue, M.D., Ph.D, Principal Investigator — Wakayama Medical University
Locations (11):
- Japan (11):
  - Kansai Rosai Hospital, Amagasaki, Hyogo
  - Kansai Medical University, Hirakata, Osaka
  - Hiroshima University, Hiroshima, Hiroshima
  - Nara Medical University, Kashihara, Nara
  - Kobe University, Kobe, Hyogo
  - Kyoto Prefectural University of Medicine, Kyoto
  - Nagoya University, Nagoya, Aichi
  - Hyogo College of Medicine, Nishinomiya, Hyogo
  - Osaka University, Osaka
  - Kinki University, Sayama, Osaka
  - Wakayama Medical University, Wakayama

REFERENCES:
- [Derived] Kawai M, Hirono S, Okada KI, Satoi S, Yanagimoto H, Kon M, Murakami Y, Kondo N, Sho M, Akahori T, Toyama H, Fukumoto T, Fujii T, Matsumoto I, Eguchi H, Ikoma H, Takeda Y, Fujimoto J, Yamaue H. Reinforced staplers for distal pancreatectomy. Langenbecks Arch Surg. 2017 Dec;402(8):1197-1204. doi: 10.1007/s00423-017-1634-1. Epub 2017 Nov 4. PMID 29103084